CLINICAL TRIAL: NCT03068390
Title: Rural Intervention for Caregivers' Heart Health (RICHH)
Brief Title: Rural Intervention for Caregivers' Heart Health
Acronym: RICHH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Debra Moser (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor-Investigator, Debra Moser, Sponsor/PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01NR016824 (NIH); 1R01NR016824 (NIH)
Record Dates: First submitted 2017-01-24; First posted 2017-03-01 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Risk Factor

STUDY DESIGN:
Intervention Model Description: 2 group randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RICHH Intervention (Experimental): The RICHH intervention is an educational-behavioral and counseling intervention that promotes caregivers' knowledge, skills and motivation to engage in CVD risk reduction. The intervention is delivered individually to caregivers in their homes using video-conferencing technology on mini-iPads that we provide for all participants. Participants keep the mini-iPads at the end of the study. The program consists of 12 weekly sessions [30-45 minutes] followed by 8 bi-weekly [every other week] booster sessions and 6 monthly booster sessions that will be held at the caregivers' preferred times using a video conferencing program. A cardiac psychiatric advanced practice nurse certified cognitive behavioral therapy will deliver the intervention.
  Interventions: Behavioral: RICHH Intervention
- Usual care (Active Comparator): The usual care control group will receive an attention placebo intervention in which the caregivers will receive mini-iPads loaded with Caregiver and CVD risk reduction pamphlets in PDF format along with the associated links from the American Heart Association. Because the investigators may identify CVD risk factors in baseline testing in participants who do not know they have them, it would be unethical not to provide at least usual care for these. Thus, all individuals enrolled in the study and in whom the investigators identify CVD risk factors will receive referral to a primary care provider for management of the CVD risk factors identified.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: RICHH Intervention — Whole health cardiovascular disease (CVD) self-care risk reduction intervention
  Arms: RICHH Intervention
Behavioral: Usual care — Referral to primary care provider
  Arms: Usual care

SUMMARY:
The investigators are testing a two-group, randomized, controlled trial with 280 primary caregivers of adult patients with a chronic illness to test the efficacy of the Rural Intervention for Caregivers' Heart Health (RICHH). Immediate (4-month) and long-term (12-month) effects of the RICHH intervention on CVD risk factors, self-management behaviors, and depressive symptoms will be compared to usual care. The investigators also will test the moderating effect of gender on intervention outcomes, given the many differences between male and female caregivers.

Specific Aim 1: To determine effects of the RICHH intervention on the primary outcomes of CVD risk factors (i.e., lipid profile, body mass index, and blood pressure) at 4 and 12 months.

Hypotheses 1: The intervention group will have better lipid profile, body mass index, and blood pressure outcomes than the usual care group at 4 and 12 months.

Specific Aim 2: To determine effects of the RICHH intervention on self-management behaviors (i.e., diet quality, physical activity level, and self-report adherence to specific CVD health behaviors).

Hypotheses 2: The intervention group will have better diet quality, higher physical activity levels, and better adherence to specific CVD health behaviors than the usual care group at 4 and 12 months.

Specific Aim 3: To determine effects of RICHH on depressive symptoms at 4 and 12 months.

Hypotheses 3: Caregivers receiving the intervention will have lower levels of depressive symptoms than caregivers receiving usual care at 4 and 12 months.

Specific Aim 4: To evaluate whether intervention effects on outcomes will differ by caregivers' gender.

Hypotheses 4: Effects will be stronger for male compared to female caregivers at 4 and 12 months.

Impact: The proposed study will have a substantial impact on caregivers' cardiovascular health and quality of life because it will provide needed CVD risk prevention, and health promotion to rural caregivers living in distressed environments where CVD risk reduction and self-management is difficult. The intervention holds the potential to produce major improvements in health among caregivers living in rural environments in the US.

ELIGIBILITY:
Inclusion Criteria:

* primary family rural caregiver of patients with chronic illnesses
* provided care for the patient for > 6 months
* no cognitive impairment that would preclude understanding the consent process

Exclusion Criteria:

* chronic drug abuse
* current active cancer
* any physical or emotional impairment that limits participants' abilities to engage in self-management or that is likely to result in needing a caregiver in the next 12 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Lipid Profile Derived from point-of-care testing | Baseline, 4 and 12 months
  lipid profile from point-of-care testing
Change in Body Mass Index (kg/m2) calculated from height and weight | Baseline, 4 and 12 months
  body mass index calculated from height and weight
Change in Blood Pressure in mmHg | Baseline, 4 and 12 months
  blood pressure

SECONDARY OUTCOMES:
Change in Diet Quality measured by the Food Frequency Questionnaire | Baseline, 4 and 12 months
  diet quality
Change in Depressive Symptoms | Baseline, 4 and 12 months
  depressive symptoms measured using PHQ-9
Change in Physical Activity Level (steps per 24 hours) measured by actigraphy | Baseline, 4 and 12 months
  physical activity levels assessed using Withings actigraph
Change in Adherence measured using the Specific Adherence Scale score from Medical Outcomes Study | Baseline, 4 and 12 months
  adherence using Specific Adherence Scale from Medical Outcomes Study

CONTACTS AND LOCATIONS:
Overall Officials: Debra K Moser, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No